CLINICAL TRIAL: NCT04896242
Title: Multimodal Assesment of Acute Cardiac Toxicity Induced by Thoracic Radiotherapy in Cancer Patients
Status: Completed | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Other Study IDs: 11190071
Record Dates: First submitted 2021-05-09; First posted 2021-05-21 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Radiotherapy; Complications; Cardiotoxicity; Cancer; Lung Cancer; Breast Cancer; Esophageal Cancer
MeSH Terms: conditions — Cardiotoxicity; Neoplasms; Lung Neoplasms; Breast Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate and compare the changes by two modalities: Imaging by Strain by Speckle Tracking and Magnetic Resonance versus soluble markers of cardiac dysfunction as early predictors of cardio-toxicity in cancer patients receiving low or high doses of radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 year-old patients
* With histologically confirmed thoracic cancer (breast, esophagus or lung)
* Recommendation of thoracic radiotherapy (RT) with curative intent
* With or without chemotherapy
* All patients must be able to read and understand Spanish
* All patients must sign informed consent form.

Exclusion Criteria:

* Patients with no medical records,
* Pregnant
* Previously diagnosed with severe left ventricular dysfunction or a cardiac insufficiency
* Patients with metastatic disease and indication of palliative RT
* Patients with significant comorbidities associated to a <5 year life expectancy.
* Patients previously treated with thoracic RT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cancer of the thoracic area (lung, breast, esophagus or other thoracic locations) that will receive curative radiotherapy to the thoracic region at Pontificia Universidad Católica de Chile.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Global Longitudinal Strain (Left Ventricle) | Baseline, 1 and 12 weeks after Treatment
  >5 Absolute drop or 12% Relative reduction from baseline

SECONDARY OUTCOMES:
Cardiac Magnetic Resonance Cinema Imaging | Baseline, 1 and 12 weeks after treatment
  Cinema imaging: Long axis balance, Balance 4 cameras, Short shaft full balance, Right ventricular balance
Cardiac Magnetic Resonance Anatomical Image | Baseline, 1 and 12 weeks after treatment
  Inversion recovery single shot balance 3D short axis covering the entire heart and aorta with free respiratory trigger
Cardiac Magnetic Resonance Flow Image | Baseline, 1 and 12 weeks after treatment
  2D outflow tract of the aorta 2D pulmonary artery outflow tract
Cardiac Magnetic Resonance Quantitative Image | Baseline, 1 and 12 weeks after treatment
  T1 map short axis apical section T1 map short axis medial section T1 map short axis basal section
  T2 map short axis apical section T2 map short axis medial section T2 map short axis basal section

OTHER OUTCOMES:
High-sensitivity Cardiac Troponin-T | Baseline, 1 and 12 weeks after treatment
  Troponin rises >99%th percentile of the upper reference limit
N-Terminal pro-Brain Natriuretic Peptide | Baseline, 1 and 12 weeks after treatment
  N-Terminal pro-Brain Natriuretic Peptide, rises >99%th percentile of the upper reference limit
Circulating Endothelial Cells | Baseline, 1 and 12 weeks after treatment
  Number of Circulating Endothelial Cells

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Merino Lara, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Pontificia Universidad Catolica de Chile, Santiago, Santiago Metropolitan, Chile